CLINICAL TRIAL: NCT04634799
Title: Study to AntagOnize Plasminogen Activator Inhibitor-1 in Severe COVID-19 (STOP Severe COVID-19)
Brief Title: Study to AntagOnize Plasminogen Activator Inhibitor-1 in Severe COVID-19
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Enrollment challenges; new batch of drug is being manufactured and there may be additional impetus to reactivate after the analogous Phase 2 study in Japan is completed and those results are made available
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Sanjiv Shah, Director of Research, Bluhm Cardiovascular Institute, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STU00213262
Record Dates: First submitted 2020-11-17; First posted 2020-11-18 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Covid19
Keywords: PAI-1; TM5614; Plasminogen Activator Inhibitor
MeSH Terms: conditions — COVID-19 | interventions — Plasminogen Activator Inhibitor 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: double-blind, randomized (1:1)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- TM5614 (Active Comparator): TM5614 30 mg tablets. 6 tablets (180 mg) taken by mouth, once daily for up to 7 days
  Interventions: Drug: TM5614
- Placebo (Placebo Comparator): Placebo tablets. 6 tablets taken by mouth, once daily for up to 7 days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: TM5614 — TM5614 is provided in 30 mg tablets and 6 tablets (180 mg) will be taken in the evening for up to 7 days.
  Other Names: Plasminogen activator inhibitor-1 (PAI-1)
  Arms: TM5614
Other: Placebo — Matching placebo will be provided and participants will take 6 tablets in the evening for up to 7 days.
  Other Names: TM5614 Placebo
  Arms: Placebo

SUMMARY:
This is a single-center, randomized double blind placebo controlled trial to evaluate the efficacy and safety of novel PAI-1 inhibitor (TM5614) for high-risk patients hospitalized with severe COVID-19 at Northwestern Memorial Hospital. The patients will be randomized in a 1:1 ratio to receive standard of care plus TM5614 or standard of care plus placebo.

DETAILED DESCRIPTION:
This project will evaluate the efficacy and safety of a novel small molecule therapy targeting PAI-1 (TM5614) for patients with severe COVID-19. This is a randomized (1:1), double-blinded trial that will enroll adult patients (> 65 years OR <65 years with at least one major cardiometabolic comorbidity [diabetes, hypertension, or cardiovascular disease]) with COVID-19 requiring supplemental oxygen. The study intervention will be a small molecule inhibitor of PAI-1, TM5614, up to 180 mg, compared to matching placebo for up to 7 days.

Research blood samples for PAI-1 and C-reactive protein (CRP) will be collected at time of enrollment, 48 hours after 1st dose of medication and at day 7 or discharge, whichever comes first.

These objectives will allow for the planning of subsequent phase 3 study, and strengthen implementation of a multi-center randomized trial should this study confirm safety, and suggest efficacy of therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥65 years old or < 65 years old AND at least one major cardiometabolic comorbidity (diabetes, hypertension, or cardiovascular disease)
2. Established diagnosis of COVID-19 as evidenced by a positive nasopharyngeal or bronchoalveolar lavage viral PCR for SARS-CoV2
3. Requiring supplemental oxygen

Exclusion Criteria:

1. Age <18 years old
2. Pregnancy or breast-feeding
3. Known contraindication to tissue plasminogen activator (tPA), including

   1. Active internal bleeding
   2. History of cerebrovascular accident
   3. Recent intracranial or intraspinal surgery or trauma
   4. Intracranial neoplasm, arteriovenous malformation or aneurysm
   5. Known bleeding diathesis
   6. Severe uncontrolled hypertension (SBP>200 persistently >12 hours)
4. Currently receiving therapeutic dose anticoagulation (specifically will exclude those with potential drug-drug interaction such as heparin, apixaban, warfarin)
5. Platelets <50,000
6. Hematocrit <30%
7. Not hemodynamically stable in the preceding 4 hours (symptomatic hypotension or systolic BP <95 mmHg at 2 out of 3 measurements)
8. Concomitant illness, physical impairment or mental condition which in the opinion of the study team / primary care physician could interfere with the conduct of the study including outcome assessment
9. Other patient characteristics (not thought to be related to COVID-19) that portend a very poor prognosis (e.g., severe liver failure, metastatic malignancy)
10. Participation in a concurrent interventional medical investigation or pharmacologic clinical trial. Patients in observational, natural history or epidemiological studies not involving an intervention are eligible.
11. Participant's responsible attending physician believes it is not appropriate for participant to participate in the study.
12. Inability or unwillingness to provide written informed consent
13. Involvement in the planning and/or conduct of the study
14. Previous randomization in the present study
15. Unable to complete study procedures.
16. Patients with active venothromboembolic disease
17. Patients who are receiving other investigational agents for COVID-19.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2025-04-23 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Clinical improvement | 7 Days
  Change of at least 2 points in the NIAID-defined ordinal scale (higher scores indicate improved outcome),:
  1. Death
  2. Hospitalized, receiving invasive mechanical ventilation or ECMO
  3. Hospitalized, receiving noninvasive ventilation or high-flow oxygen devices
  4. Hospitalized, requiring low-flow supplemental oxygen
  5. Hospitalized, not requiring supplemental oxygen but receiving ongoing medical care (related or not related to Covid-19)
  6. Hospitalized, requiring neither supplemental oxygen nor ongoing medical care (other than that specified in the protocol)
  7. Not hospitalized

SECONDARY OUTCOMES:
Sequential organ failure assessment (SOFA) score change | 7 Days
  Change in degree of organ dysfunction as defined by the Sequential Organ Failure Assessment (SOFA) Score.
  The SOFA score ranges from 0 to 24 (higher scores indicate more severe organ failure), with 0 to 4 points assigned for each of 6 organ dysfunctions (ie, central nervous system, cardiovascular, respiratory, renal, coagulation, and liver).
PAI-1 Levels | 48 hours
  Change in circulating levels
Ventilator free days | 14 days
  For subjects who received mechanical ventilation, total number of days the subject was not on mechanical or non invasive mechanical ventilation while in the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Sanjiv Shah, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chang D, Lin M, Wei L, Xie L, Zhu G, Dela Cruz CS, Sharma L. Epidemiologic and Clinical Characteristics of Novel Coronavirus Infections Involving 13 Patients Outside Wuhan, China. JAMA. 2020 Mar 17;323(11):1092-1093. doi: 10.1001/jama.2020.1623. PMID 32031568
- [Background] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Liu YC, Liao CH, Chang CF, Chou CC, Lin YR. A Locally Transmitted Case of SARS-CoV-2 Infection in Taiwan. N Engl J Med. 2020 Mar 12;382(11):1070-1072. doi: 10.1056/NEJMc2001573. Epub 2020 Feb 12. No abstract available. PMID 32050059